CLINICAL TRIAL: NCT01987336
Title: A Prospective Anaylsis of Biofilm in Urinary Catheters Study
Brief Title: A Prospective Analysis of Biofilm in Urinary Catheters Study
Status: Completed | Type: Observational
Sponsor: Southwest Regional Wound Care Center (Other)
Responsible Party: Sponsor
Other Study IDs: 56-RW-022
Record Dates: First submitted 2013-03-04; First posted 2013-11-19 (Estimated); Last update posted 2015-12-11 (Estimated); Status verified 2015-12

CONDITIONS: Urinary Incontinence
Keywords: Standard Foley Catheter
MeSH Terms: conditions — Urinary Incontinence

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — A 30cc urine sample would also be collected, along with the used catheter. The molecular evaluation will be looking specifically at the biofilm accumulated on the catheter surface. The technologies to be used are proteomics, metabolomics and metagenomics.
Oversight: Data Monitoring Committee: No

SUMMARY:
To analyze biofilm obtained from at least 10 Subjects who have an indwelling catheter. A 30cc urine sample would also be collected from the same subject, and analyzed.

DETAILED DESCRIPTION:
After obtaining informed consent, concurrent with the changing of the Foley catheter in the clinic, would be obtaining a 30 cc. sample of urine which would also be fast frozen and stored in a -81 degree freezer until shipped to the Venter clinic on dry ice.

ELIGIBILITY:
Inclusion Criteria:

1. Subject must be 18 years of age.
2. Subject is attending weekly office visits at SW Wound Care Center as an out- patient.
3. Subject must have an indwelling Foley catheter.
4. Subject is informed about the trial, understands its nature of the study and provides written informed consent prior to study enrollment.
5. Subject is willing and able to comply with all specified care and visit requirements.

Exclusion Criteria:

1. Subject refuses to participate in the study. 2. Subject is expected to be non-compliant. 3. Subject is a resident in a nursing home, or institutionalized. 4. Subject is pregnant. 5. Subject has a Legally Authorized Representative

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Subjects who require a standard foley catheter.
Sampling Method: Non-Probability Sample
Enrollment: 9 (Actual)
Dates: Start 2013-03; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
To analyze biofilm obtained from at least 10 Subjects who have an indwelling catheter. | Over a period of 20 weeks
  the proteomics, metabolomics and metagenomics ("omics") data will be analyzed and integrated in order to understand the microbial population dynamics and the interactions with the human subject host responses which may include antibacterial defenses, local inflammation, immune tolerance towards bacteria

CONTACTS AND LOCATIONS:
Overall Officials: Randall Wolcott, M.D., Principal Investigator — Southwest Regional Wound Care Center
Locations (1):
- Southwest Regional Wound Care Center, Lubbock, Texas, United States